CLINICAL TRIAL: NCT05259241
Title: Correlation Between ACT anD APTT During Transcatheter Aortic Valve Implantation and Chronic Total Occlusion Percutaneous Coronary Interventions
Brief Title: ADAPT Transcatheter Aortic Valve Intervention (TAVI & Chronic Total Occlusion Percutaneous Coronary Intervention (CTO PCI)
Acronym: ADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Clinical director of Interventional cardiology, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC-2020-0375
Record Dates: First submitted 2021-09-21; First posted 2022-02-28 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Transcatheter Aortic Valve Replacement; Percutaneous Coronary Intervention
Keywords: ACT; APTT

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): Cohort A: patients undergoing TAVR to evaluate which point-of-care test (ACT or aPTT) gives the best correlation with the coagulation status
  Cohort B: patients undergoing PCI to evaluate which point-of-care test (ACT or aPTT) gives the best correlation with the coagulation status
  Interventions: Diagnostic Test: activated partial thrombin time

INTERVENTIONS:
Diagnostic Test: activated partial thrombin time — This study aims to find which the point-of-care test (ACT or APTT) has the best correlation with the coagulation status during transcatheter cardiac interventions (either TAVR or PCI)
  Other Names: activated clotting time

SUMMARY:
Rationale: The choice of antithrombotic regimen during TAVI and CTO PCI includes the use of unfractionated heparin. The accuracy of ACT in this setting is disputed. ACT has never been compared to a point-of-care aPTT test for monitoring anticoagulation during percutaneous cardiac interventions.

Objective: The aim of the present study is to evaluate which point-of-care test (ACT or aPTT) gives the best correlation with the coagulation status in patients, defined with the anti-Xa measurement.

Study design: A Single-center, prospective, observational study Study population: patients undergoing TAVI (Cohort A) or CTO PCI (Cohort B) in the Erasmus University Medical Center

Main study parameters/endpoints: The main study endpoints are the correlation between the ACT and APTT point-of-care- tests and the coagulation status, defined as the laboratory anti-Xa measurement.

DETAILED DESCRIPTION:
The choice of antithrombotic regimen during TAVI and CTO PCI includes the use of unfractionated heparin. Heparin is the preferred anticoagulant drug in these percutaneous cardiac interventions aiming for an Activated Clotting Time (ACT) > 200sec or 250seconds depending on the procedure. Heparin has a short half-life time and can be neutralized by protamine.

Monitoring the use of unfractionated heparin during TAVI and PCI can be performed with several measurements, like the ACT and aPTT. To measure ACT, an activator is mixed with whole blood to provide a timing of haemostasis. aPTT is a plasma test in which a surface activator is used to measure the time it takes to form a fibrin clot. In nearly every center ACT is the preferred method because of its ease of use and the assumed reliability. ACT-guided heparin regime during TAVI seems effective in minimizing major bleeding events.

There are limited studies focussing on the difference between ACT- and aPTT measurements. The studies which investigated this difference are merely done in patients with continuous heparin infusions, for example in the setting of extracorporeal membrane oxygenation(ECMO). These studies suggest that there is a better correlation between aPTT and dosage heparin than between ACT and heparin. Also, the correlation between ACT and aPTT seems poor.

The accuracy and correlation of ACT with a point-of-care aPTT test for monitoring the anticoagulation effect of unfractionated heparin has so far not been done in the setting of percutaneous interventions. TAVI requires large bore arterial access and is associated with a relevant frequency of access site related bleeding and vascular complications. CTO procedures often require dual arterial access and the use of different strategies with multiple wires which increases the prevalence of vascular complications, including pericardial effusion.

Precise knowledge of actual anticoagulation status during an invasive procedure and at the time of access site closure may affect the incidence of TAVI and CTO PCI related bleeding complications.

Therefore, the aim of the present study is to evaluate which point-of-care test (ACT or aPTT) gives the best correlation with the coagulation status in patients during TAVI and CTO PCI.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a TAVI-procedure
* All patients undergoing a CTO PCI procedure

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between the ACT point-of-care test with the Anti-Xa-activity measurement). | 30 minutes after heparin bolus
  The anti-Xa-measurement(in IU/mL) is defined as the reference for the coagulation status. In this study, we measure the point-of-care ACT measurement(in milliseconds) and the anti-Xa measurement 30 minutes after the heparin bolus to determine the correlation.
The correlation between the APTT point-of-care test with the coagulation status(Anti-Xa-measurement). | 30 minutes after heparin bolus
  The anti-Xa-measurement(in IU/mL) is defined as the reference for the coagulation status. In this study, we measure the point-of-care APTT measurement(in milliseconds) and the anti-Xa measurement 30 minutes after the heparin bolus to determine the correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided